CLINICAL TRIAL: NCT00544375
Title: Non-Invasive Measurements of Anemia and Physiologic Tissue Response to Blood Transfusions in Very Low Birth Weight Infants Using Quantitative Near-Infrared Spectroscopy
Brief Title: Measurements of Anemia and Physiologic Tissue Response to Blood Transfusions in VLBW Infants Using Quantitative NIRS
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Feizal Waffarn, M.D, University of California, Irvine
Other Study IDs: 20012011
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Infant Development

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neonatal Tissues: Optical measurement neonatal tissues
  Interventions: Device: Optical measurement

INTERVENTIONS:
Device: Optical measurement — Optical measurement neonatal tissues

SUMMARY:
The study quantified functional measures of red blood cell mass and oxygen in neonatal tissues using a non-invasive optical technique: near infrared optical spectroscopy . The study will determine the absolute concentrations of deoxygenated and oxygenated hemoglobin and calculate the tissue hemoglobin saturation and total hemoglobin concentration in viv. Near infrared optical spectroscopy technique use to assessing and defining tissue status in the anemic state and the tissue's response to transfusions, as well as in monitoring hemoglobin and hematocrit without pain or loss of blood.

DETAILED DESCRIPTION:
Near infrared optical spectroscopy measurements will be conducted on the muscle, on the upper leg,arm or on the back, abdomen and the head. The actual location will depend upon the neonate position and size. A small soft plastic optical fibers probe will be placed to the select study areas and thhe time of the measurement will not exceed 1 hour.

NIRS measurements of hemoglobin and hemoglobin saturation in tissues before and after red-cell transfusions in VLBW infants will determine the true effect of the transfusions, and develop more substantial guidelines regarding indications for transfusion. The accuracy of conventional (invasive) measurements of Hb and Hct could be comparison with results from the NIRS technique and clinical usefulness of the NIRS technique could be evaluated by comparison with trends in conventionally measured values taking fluid status into account.

Near-infrared light does not ionize biological tissue and poses no significant health risk. Since water absorption is low within this spectral range, local heating of the tissue is also minimal. Burns and heat damage to the neonate are highly unlikely.

ELIGIBILITY:
Inclusion Criteria:

* infants weighing less than 1500 grams at birth
* infants receiving at least one packed red blood cell transfusion

Exclusion Criteria:

* neonates who are too unstable as determined by the clinicians for additional human contact

Ages: 1 Minute to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2002-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Infant tissue's response to transfusions | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Feizal Waffarn, M.D, Principal Investigator — Beckman Laser Institute University of California Irvine; Bruce Tromberg, PhD, Study Director — Beckman Laser Institute University of California Irvine
Locations (1):
- Neonatal Intensive Care Unit, University of California Irvine, Orange, California, United States